CLINICAL TRIAL: NCT00416156
Title: Effect of Weight Reduction on Inflammatory Markers and Genes Expression in Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: TCVGH 05082
Record Dates: First submitted 2006-12-25; First posted 2006-12-27 (Estimated); Last update posted 2006-12-27 (Estimated); Status verified 2006-12

CONDITIONS: Obesity; Inflammation
Keywords: Obesity; Inflammation
MeSH Terms: conditions — Obesity; Inflammation

INTERVENTIONS:
Behavioral: Lifestyle modification

SUMMARY:
To investigate whether weight reduction by life style modification for 12 weeks will improve circulating inflammatory markers, adipocytokines as well as gene expression of proinflammatory protein obtained from circulating monocytes from obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* Nondiabetes obese individuals with BMI greater than 27 kgs/m2

Exclusion Criteria:

* Diabetes
* Abnormal hepatic, renal and cardiac function

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2005-05; Study Completion 2005-11

PRIMARY OUTCOMES:
Inflammatory responses after weight reduction

SECONDARY OUTCOMES:
BMI
Circulating inflammatory markers
Adipocytokines
Gene Expression from mononuclear cells

CONTACTS AND LOCATIONS:
Overall Officials: Wayne H Sheu, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan